CLINICAL TRIAL: NCT01847313
Title: Phase 3 Study of the Effect of Glucagon-like-peptide 1 (GLP-1) Receptor Agonism on Renal Outcomes in Humans With Diabetic Kidney Disease
Brief Title: The Effect of Glucagon-like-peptide 1 (GLP-1) Receptor Agonism on Diabetic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karl Neff (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Sponsor-Investigator, Karl Neff, Clinical Research Fellow, University College Dublin
Organization: University College Dublin (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLP-1-2012-01
Record Dates: First submitted 2013-04-29; First posted 2013-05-06 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-02-08 (Actual); Status verified 2018-09

CONDITIONS: Diabetic Kidney Disease
Keywords: kidney; diabetes; glp-1
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Active Comparator): Liraglutide 0.6 mg daily
  Interventions: Drug: Liraglutide
- Control (No Intervention): Standard diabetes care including renin angiotensin aldosterone system inhibitor or antagonist

INTERVENTIONS:
Drug: Liraglutide — Daily administration of liraglutide for 6 months
  Other Names: Glucagon like peptide 1 receptor agonist; NN2211
  Arms: Liraglutide

SUMMARY:
Diabetic kidney disease (DKD) is a devastating complication of diabetes, that in it's worst form, can lead to early cardiovascular death or kidney failure. A group of medicines used to treat diabetes, glucagon-like-peptide-1 analogues (GLP-1), may be able to protect people with diabetes from DKD by reducing inflammation in the kidney. This study aims to test this theory by studying the effect of GLP-1 on kidney function in people with diabetes.

To understand how GLP-1 can affect inflammation, the investigators will give a GLP-1 treatment (Liraglutide) to people with DKD and monitor the effect on inflammation and kidney function using blood and urine tests. The investigators will compare these results to patients with DKD who do not receive GLP-1 treatment.

If GLP-1 proves to be effective in reducing inflammation and improving kidney function, then it could be developed as a viable new treatment for people with DKD, and may significantly reduce the disease burden, or the risk of DKD, in people with diabetes. This would be a major advance in the treatment of DKD.

DETAILED DESCRIPTION:
A randomised controlled trial for patients with microalbuminuria and type 2 diabetes. Treatment is 0.6mg of liraglutide and is compared to standard care. Treatment duration is 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with a HbA1c of 42-75mmol/mol (6-9%DCCT)
* Male or female aged above 30 years
* Have a negative pregnancy test at screening (women of child bearing potential only)
* Body mass index (BMI) of 25kg/m2 or greater
* On a renin-angiotensin system antagonist, at a stable dose, for at least 8 weeks before inclusion into the study
* Established microalbuminuria
* Estimated glomerular filtration rate (eGFR) 30ml/min/1.73m2 or above by Modification of Diet in Renal Disease (MDRD) formula

Exclusion Criteria:

* Patients with any cognitive impediment that preclude the patient from giving free and informed consent
* Patients on dipeptidyl peptidase 4 inhibitors or thiazolidinedione treatment
* Patients with stage 4-5 renal disease, defined as an eGFR of 30ml/min/1.73m2 or less
* Patients who have used a GLP-1 agent in the last 6 months
* Female patients of child bearing potential who are pregnant, breastfeeding, or unwilling to practice an acceptable barrier and/or hormonal method of contraception or abstinence during participation in the study
* Previous pancreatitis
* Hypersensitivity to GLP-1 analogues
* Proliferative diabetic retinopathy
* Any other contraindications, as per the SmPC for liraglutide
* Patients with any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the dosing requirements
* Concurrent treatment with an investigational drug or participation in another clinical trial
* Use of an investigational drug within 4 weeks or 5 half-lives, whichever is longer, preceding the first dose of investigational medicinal product

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carel le Roux, MBBS PhD, Study Director — University College Dublin
Locations (1):
- St Vincent's Healthcare Group, Dublin, Ireland

REFERENCES:
- [Background] Fenske WK, Dubb S, Bueter M, Seyfried F, Patel K, Tam FW, Frankel AH, le Roux CW. Effect of bariatric surgery-induced weight loss on renal and systemic inflammation and blood pressure: a 12-month prospective study. Surg Obes Relat Dis. 2013 Jul-Aug;9(4):559-68. doi: 10.1016/j.soard.2012.03.009. Epub 2012 Apr 10. PMID 22608055
- [Background] Miras AD, Chuah LL, Lascaratos G, Faruq S, Mohite AA, Shah PR, Gill M, Jackson SN, Johnston DG, Olbers T, le Roux CW. Bariatric surgery does not exacerbate and may be beneficial for the microvascular complications of type 2 diabetes. Diabetes Care. 2012 Dec;35(12):e81. doi: 10.2337/dc11-2353. No abstract available. PMID 23173142
- [Background] Meguid El Nahas A, Bello AK. Chronic kidney disease: the global challenge. Lancet. 2005 Jan 22-28;365(9456):331-40. doi: 10.1016/S0140-6736(05)17789-7. PMID 15664230
- [Background] Navarro-Gonzalez JF, Mora-Fernandez C, Muros de Fuentes M, Garcia-Perez J. Inflammatory molecules and pathways in the pathogenesis of diabetic nephropathy. Nat Rev Nephrol. 2011 Jun;7(6):327-40. doi: 10.1038/nrneph.2011.51. Epub 2011 May 3. PMID 21537349
- [Background] Lim AK, Tesch GH. Inflammation in diabetic nephropathy. Mediators Inflamm. 2012;2012:146154. doi: 10.1155/2012/146154. Epub 2012 Aug 21. PMID 22969168
- [Background] Shyangdan DS, Royle P, Clar C, Sharma P, Waugh N, Snaith A. Glucagon-like peptide analogues for type 2 diabetes mellitus. Cochrane Database Syst Rev. 2011 Oct 5;2011(10):CD006423. doi: 10.1002/14651858.CD006423.pub2. PMID 21975753
- [Background] Hogan AE, Tobin AM, Ahern T, Corrigan MA, Gaoatswe G, Jackson R, O'Reilly V, Lynch L, Doherty DG, Moynagh PN, Kirby B, O'Connell J, O'Shea D. Glucagon-like peptide-1 (GLP-1) and the regulation of human invariant natural killer T cells: lessons from obesity, diabetes and psoriasis. Diabetologia. 2011 Nov;54(11):2745-54. doi: 10.1007/s00125-011-2232-3. Epub 2011 Jul 9. PMID 21744074
- [Background] Lynch LA, O'Connell JM, Kwasnik AK, Cawood TJ, O'Farrelly C, O'Shea DB. Are natural killer cells protecting the metabolically healthy obese patient? Obesity (Silver Spring). 2009 Mar;17(3):601-5. doi: 10.1038/oby.2008.565. Epub 2008 Dec 18. PMID 19238145
- [Background] Lynch L, O'Shea D, Winter DC, Geoghegan J, Doherty DG, O'Farrelly C. Invariant NKT cells and CD1d(+) cells amass in human omentum and are depleted in patients with cancer and obesity. Eur J Immunol. 2009 Jul;39(7):1893-901. doi: 10.1002/eji.200939349. PMID 19585513
- [Background] Chow FY, Nikolic-Paterson DJ, Ozols E, Atkins RC, Rollin BJ, Tesch GH. Monocyte chemoattractant protein-1 promotes the development of diabetic renal injury in streptozotocin-treated mice. Kidney Int. 2006 Jan;69(1):73-80. doi: 10.1038/sj.ki.5000014. PMID 16374426
- [Background] Chow F, Ozols E, Nikolic-Paterson DJ, Atkins RC, Tesch GH. Macrophages in mouse type 2 diabetic nephropathy: correlation with diabetic state and progressive renal injury. Kidney Int. 2004 Jan;65(1):116-28. doi: 10.1111/j.1523-1755.2004.00367.x. PMID 14675042
- [Background] Kanamori H, Matsubara T, Mima A, Sumi E, Nagai K, Takahashi T, Abe H, Iehara N, Fukatsu A, Okamoto H, Kita T, Doi T, Arai H. Inhibition of MCP-1/CCR2 pathway ameliorates the development of diabetic nephropathy. Biochem Biophys Res Commun. 2007 Sep 7;360(4):772-7. doi: 10.1016/j.bbrc.2007.06.148. Epub 2007 Jul 6. PMID 17631861
- [Background] Tarabra E, Giunti S, Barutta F, Salvidio G, Burt D, Deferrari G, Gambino R, Vergola D, Pinach S, Perin PC, Camussi G, Gruden G. Effect of the monocyte chemoattractant protein-1/CC chemokine receptor 2 system on nephrin expression in streptozotocin-treated mice and human cultured podocytes. Diabetes. 2009 Sep;58(9):2109-18. doi: 10.2337/db08-0895. Epub 2009 Jul 8. PMID 19587356
- [Background] Navarro JF, Milena FJ, Mora C, Leon C, Garcia J. Renal pro-inflammatory cytokine gene expression in diabetic nephropathy: effect of angiotensin-converting enzyme inhibition and pentoxifylline administration. Am J Nephrol. 2006;26(6):562-70. doi: 10.1159/000098004. Epub 2006 Dec 13. PMID 17167242
- [Background] Yozai K, Shikata K, Sasaki M, Tone A, Ohga S, Usui H, Okada S, Wada J, Nagase R, Ogawa D, Shikata Y, Makino H. Methotrexate prevents renal injury in experimental diabetic rats via anti-inflammatory actions. J Am Soc Nephrol. 2005 Nov;16(11):3326-38. doi: 10.1681/ASN.2004111011. Epub 2005 Sep 21. PMID 16177002
- [Background] Tone A, Shikata K, Sasaki M, Ohga S, Yozai K, Nishishita S, Usui H, Nagase R, Ogawa D, Okada S, Shikata Y, Wada J, Makino H. Erythromycin ameliorates renal injury via anti-inflammatory effects in experimental diabetic rats. Diabetologia. 2005 Nov;48(11):2402-11. doi: 10.1007/s00125-005-1945-6. Epub 2005 Oct 18. PMID 16231067
- [Background] Blandino-Rosano M, Perez-Arana G, Mellado-Gil JM, Segundo C, Aguilar-Diosdado M. Anti-proliferative effect of pro-inflammatory cytokines in cultured beta cells is associated with extracellular signal-regulated kinase 1/2 pathway inhibition: protective role of glucagon-like peptide -1. J Mol Endocrinol. 2008 Jul;41(1):35-44. doi: 10.1677/JME-07-0154. Epub 2008 May 16. PMID 18487229
- [Background] Kodera R, Shikata K, Kataoka HU, Takatsuka T, Miyamoto S, Sasaki M, Kajitani N, Nishishita S, Sarai K, Hirota D, Sato C, Ogawa D, Makino H. Glucagon-like peptide-1 receptor agonist ameliorates renal injury through its anti-inflammatory action without lowering blood glucose level in a rat model of type 1 diabetes. Diabetologia. 2011 Apr;54(4):965-78. doi: 10.1007/s00125-010-2028-x. Epub 2011 Jan 21. PMID 21253697
- [Background] Ahern T, Tobin AM, Corrigan M, Hogan A, Sweeney C, Kirby B, O'Shea D. Glucagon-like peptide-1 analogue therapy for psoriasis patients with obesity and type 2 diabetes: a prospective cohort study. J Eur Acad Dermatol Venereol. 2013 Nov;27(11):1440-3. doi: 10.1111/j.1468-3083.2012.04609.x. Epub 2012 Jun 13. PMID 22691169
- [Background] Hattori S. Sitagliptin reduces albuminuria in patients with type 2 diabetes. Endocr J. 2011;58(1):69-73. doi: 10.1507/endocrj.k10e-382. Epub 2010 Dec 28. PMID 21206136
- [Background] Cummings BP, Stanhope KL, Graham JL, Baskin DG, Griffen SC, Nilsson C, Sams A, Knudsen LB, Raun K, Havel PJ. Chronic administration of the glucagon-like peptide-1 analog, liraglutide, delays the onset of diabetes and lowers triglycerides in UCD-T2DM rats. Diabetes. 2010 Oct;59(10):2653-61. doi: 10.2337/db09-1564. Epub 2010 Jul 9. PMID 20622169
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Pinkney J, Fox T, Ranganath L. Selecting GLP-1 agonists in the management of type 2 diabetes: differential pharmacology and therapeutic benefits of liraglutide and exenatide. Ther Clin Risk Manag. 2010 Sep 7;6:401-11. doi: 10.2147/tcrm.s7313. PMID 20856686
- [Background] Jacobsen LV, Hindsberger C, Robson R, Zdravkovic M. Effect of renal impairment on the pharmacokinetics of the GLP-1 analogue liraglutide. Br J Clin Pharmacol. 2009 Dec;68(6):898-905. doi: 10.1111/j.1365-2125.2009.03536.x. PMID 20002084
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from St Vincent's University Hospital, Dublin, Ireland
Groups:
- Liraglutide: Liraglutide 0.6 mg daily administration for 6 months
Period: Overall Study
Arm/Group | Liraglutide | Control
Started | 10 | 10
Completed | 10 | 8
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7) | 64 (10) | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 7 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Ireland | 10 | 10 | 20
BMI [Mean (Standard Deviation); unit: kg/m2] | 30 (5) | 34 (4) | 32 (5)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 8 (1) | 9 (2) | 9 (2)
HbA1c [Mean (Standard Deviation); unit: mmol/mol] | 53 (7) | 52 (7) | 53 (7)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 136 (14) | 140 (20) | 138 (17)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 82 (8) | 81 (12) | 81 (10)
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: ml/min/1.73m2] | 69 (7) | 79 (11) | 74 (10)
Urinary albumin excretion rate [Mean (Standard Deviation); unit: µg/min] — Albuminuria as Measured by 24 Hour Albumin Excretion Rate
  µg/min | 106.9 (109.5) | 122.8 (142.1) | 114.9 (123.7)
MCP-1:Creatinine Ratio in Urine [Mean (Standard Deviation); unit: ng/mmol] — Spot urine sample for MCP-1 and creatinine Population: Liraglutide group contained an analytical outlier which was excluded from further analysis.
  ng/mmol
    number analyzed (Participants) | 9 | 8 | 17
    (all) | 32.8 (25.7) | 20.8 (6.0) | 27.2 (19.6)
sCD163:creatinine ratio in urine [Mean (Standard Deviation); unit: pg/mmol] — Spot urine sample for MCP-1 and creatinine Population: Baseline measure not reported for subjects that died or withdrew
  pg/mmol
    number analyzed (Participants) | 10 | 8 | 18
    (all) | 51 (60) | 37 (38) | 44 (51)
sCD163 in serum [Mean (Standard Deviation); unit: ng/ml] — Serum sample for sCD163 Population: Measure Analysis Population Description: Baseline measure not reported for subjects that died or withdrew
  ng/ml
    number analyzed (Participants) | 10 | 8 | 18
    (all) | 96 (45) | 106 (47) | 100 (45)

OUTCOME MEASURES:

1. Primary Outcome: MCP-1:Creatinine Ratio in Urine
Description: Spot urine sample for MCP-1 and creatinine
Time Frame: Up to 26 weeks
Population: Liraglutide group contained an analytical outlier which was excluded from further analysis.
Measure: Mean (Standard Deviation); unit: ng/mmol
Arm/Group | Liraglutide | Control
Number analyzed (Participants) | 9 | 8
ng/mmol | 27.9 (14.3) | 24.3 (15.4)

2. Secondary Outcome: Urine Albumin:Creatinine Ratio
Description: Spot urine sample for albumin and creatinine
Time Frame: Up to 26 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Urinary Albumin Excretion Rate
Description: Albuminuria as Measured by 24 Hour Albumin Excretion Rate
Time Frame: Up to 26 weeks
Measure: Mean (Standard Deviation); unit: µg/min
Arm/Group | Liraglutide | Control
Number analyzed (Participants) | 9 | 7
µg/min | 144.1 (232.6) | 132.4 (101.3)

4. Secondary Outcome: sCD163 in Serum
Description: Serum sample for sCD163
Time Frame: Up to 26 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Liraglutide | Control
Number analyzed (Participants) | 10 | 8
ng/ml | 82 (34) | 84 (23)

5. Secondary Outcome: sCD163:Creatinine Ratio in Urine
Description: Spot urine sample for MCP-1 and creatinine
Time Frame: Up to 26 weeks
Measure: Mean (Standard Deviation); unit: pg/mmol
Arm/Group | Liraglutide | Control
Number analyzed (Participants) | 10 | 8
pg/mmol | 27.9 (14.0) | 24.3 (15.4)

6. Other Pre Specified Outcome: Safety in All Participants as Measured by Adverse Event Rate
Description: Adverse event data collection
Time Frame: Up to 34 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Starting from the first administration of the IMP through to the End of Study Visit (30 weeks) all Adverse Event and Serious Adverse event information was collected at each visit.
Description: AEs were collected by the PI and Sub-investigators and recorded in the CRF/site file/medical record. AEs/SAEs were recorded in the CRF module for AE in verbatim terms. In case of several signs/symptoms, a single syndrome or diagnosis was recorded. In the event of an AE, investigators adjudicated whether the AE was serious, the start date, the stop date, whether the AE was related to study drug or procedure, AE-related actions taken with the study drug, the severity of the AE and outcome.
Arm/Group | Liraglutide | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/10
Other Adverse Events (participants affected / at risk) | 8/10 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=10) | Control (N=10)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1) — Exacerbation of pre-existing heart!failure
Paroxysmal atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=10) | Control (N=10)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Hypokalaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Viral illness (Infections and infestations) | 0 (0) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (7) | 1 (9)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ingrown toenail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Mouth ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Hyponatraemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No